CLINICAL TRIAL: NCT07142668
Title: The Impact of Availability of Conventional Cigarettes and LNCs in the Context of Innovative Tax Proposals
Brief Title: Effects of Tax Proposals and Cigarette Availability on Tobacco Purchasing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Roswell Park Comprehensive Cancer Center (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Stein, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VT IRB 25-612; R01CA266966 (NIH)
Record Dates: First submitted 2025-08-07; First posted 2025-08-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cigarette Smoking
Keywords: Experimental Tobacco Marketplace
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Participants will complete two control trials and one Experimental Marketplace condition, representing one of the four tax proposals. Within each tax policy group, each participant will complete five purchase scenarios in which conventional cigarettes are available and five in which conventional cigarettes are not available. In each condition, taxes will be increased proportionally across five trials to examine how cigarette purchasing and product substitution are affected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tobacco Parity (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to two control trials and the Tobacco Parity Tax condition. Tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all tobacco products are placed in the high-tax tier while products that do not contain tobacco (e.g., herbal cigarettes and nicotine-free ENDS) are placed in the medium-tax tier. Nicotine Replacement Therapy products are placed in the no-tax tier.
  Interventions: Behavioral: Tobacco Parity Tax - Normal Nicotine Cigarettes Available; Behavioral: Tobacco Parity Tax - Normal Nicotine Cigarettes Not Available
- Nicotine Content (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to two control trials and the Nicotine-Content Tax Condition. Products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, products with greater than 3 mg nicotine per single unit are placed in the high-tax tier, products with 0.6-3.0 mg/unit in the medium-tax tier, and those with 0.5 mg/unit or less in the no-tax tier.
  Interventions: Behavioral: Nicotine Content Tax - Normal Nicotine Cigarettes Available; Behavioral: Nicotine Content Tax - Normal Nicotine Cigarettes Not Available
- Harm Reduction (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to two control trials and the Harm Reduction Tax Condition. Tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all combustible products with high abuse liability are placed in the high-tax tier. All non-combustible products or combustible products with low abuse liability are placed in the medium-tax tier. Nicotine Replacement Therapy products are placed in the no-tax tier.
  Interventions: Behavioral: Harm Reduction Tax - Normal Nicotine Cigarettes Available; Behavioral: Harm Reduction Tax - Normal Nicotine Cigarettes Not Available
- Modified Risk Tobacco Products (MRTP) (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to two control trials and the Modified Risk Tobacco Products tax condition. Tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all non-MRTP tobacco products are placed in the high-tax tier, MRTPs are placed in the medium-tax tier, and Nicotine Replacement Therapy products are placed in the no-tax tier.
  Interventions: Behavioral: Modified Risk Tobacco Product Tax - Normal Nicotine Cigarettes Available; Behavioral: Modified Risk Tobacco Product Tax - Normal Nicotine Cigarettes Not Available

INTERVENTIONS:
Behavioral: Harm Reduction Tax - Normal Nicotine Cigarettes Available — In the Harm Reduction Tax Condition, tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. All combustible products with high abuse liability are placed in the high-tax tier. All non-combustible products or combustible products with low abuse liability are placed in the medium-tax tier. Nicotine Replacement Therapy products are placed in the no-tax tier. The participant's preferred normal-nicotine content cigarettes are available in the marketplace. Participants complete two trials with all products offered at market price, and five trials with prices for each product increasing proportionally to tax tier.
  Arms: Harm Reduction
Behavioral: Harm Reduction Tax - Normal Nicotine Cigarettes Not Available — In the Harm Reduction Tax Condition, tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. All combustible products with high abuse liability are placed in the high-tax tier. All non-combustible products or combustible products with low abuse liability are placed in the medium-tax tier. Nicotine Replacement Therapy products are placed in the no-tax tier. The participant's preferred normal-nicotine content cigarettes are NOT available in the marketplace. Participants complete two trials with all products offered at market price, and five trials with prices for each product increasing proportionally to tax tier.
  Arms: Harm Reduction
Behavioral: Modified Risk Tobacco Product Tax - Normal Nicotine Cigarettes Available — In the Modified Risk Tobacco Products tax condition, tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all non-MRTP tobacco products are placed in the high-tax tier, MRTPs are placed in the medium-tax tier, and Nicotine Replacement Therapy products are placed in the no-tax tier. The participant's preferred normal-nicotine content cigarettes are available in the marketplace. Participants complete two trials with all products offered at market price, and five trials with prices for each product increasing proportionally to tax tier.
  Arms: Modified Risk Tobacco Products (MRTP)
Behavioral: Modified Risk Tobacco Product Tax - Normal Nicotine Cigarettes Not Available — In the Modified Risk Tobacco Products tax condition, tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all non-MRTP tobacco products are placed in the high-tax tier, MRTPs are placed in the medium-tax tier, and Nicotine Replacement Therapy products are placed in the no-tax tier. The participant's preferred normal-nicotine content cigarettes are NOT available in the marketplace. Participants complete two trials with all products offered at market price, and five trials with prices for each product increasing proportionally to tax tier.
  Arms: Modified Risk Tobacco Products (MRTP)
Behavioral: Nicotine Content Tax - Normal Nicotine Cigarettes Available — In the Nicotine-Content Tax Condition, products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, products with greater than 3 mg nicotine per single unit are placed in the high-tax tier, products with 0.6-3.0 mg/unit in the medium-tax tier, and those with 0.5 mg/unit or less in the no-tax tier. The participant's preferred normal-nicotine content cigarettes are available in the marketplace. Participants complete two trials with all products offered at market price, and five trials with prices for each product increasing proportionally to tax tier.
  Arms: Nicotine Content
Behavioral: Nicotine Content Tax - Normal Nicotine Cigarettes Not Available — In the Nicotine-Content Tax Condition, products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, products with greater than 3 mg nicotine per single unit are placed in the high-tax tier, products with 0.6-3.0 mg/unit in the medium-tax tier, and those with 0.5 mg/unit or less in the no-tax tier. The participant's preferred normal-nicotine content cigarettes are NOT available in the marketplace. Participants complete two trials with all products offered at market price, and five trials with prices for each product increasing proportionally to tax tier.
  Arms: Nicotine Content
Behavioral: Tobacco Parity Tax - Normal Nicotine Cigarettes Available — In the Tobacco Parity Tax condition, tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all tobacco products are placed in the high-tax tier while products that do not contain tobacco (e.g., herbal cigarettes and nicotine-free ENDS) are placed in the medium-tax tier. Nicotine Replacement Therapy products are placed in the no-tax tier. The participant's preferred normal-nicotine content cigarettes are available in the marketplace. Participants complete two trials with all products offered at market price, and five trials with prices for each product increasing proportionally to tax tier.
  Arms: Tobacco Parity
Behavioral: Tobacco Parity Tax - Normal Nicotine Cigarettes Not Available — In the Tobacco Parity Tax condition, tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all tobacco products are placed in the high-tax tier while products that do not contain tobacco (e.g., herbal cigarettes and nicotine-free ENDS) are placed in the medium-tax tier. Nicotine Replacement Therapy products are placed in the no-tax tier. The participant's preferred normal-nicotine content cigarettes are NOT available in the marketplace. Participants complete two trials with all products offered at market price, and five trials with prices for each product increasing proportionally to tax tier.
  Arms: Tobacco Parity

SUMMARY:
This study will investigate the effects of normal-nicotine versus low-nicotine cigarette availability in the context of four tax proposals (Tobacco Parity, Nicotine-Content, Harm-Reduction, and Modified Risk Tobacco Product-based taxes) on tobacco product purchasing patterns in a virtual marketplace.

DETAILED DESCRIPTION:
In a within/between subjects design, the investigators will use an Experimental Tobacco Marketplace (ETM) to systematically impose four innovative tobacco/nicotine tax proposals (Tobacco Parity, Nicotine-Content, Harm-Reduction, and Modified Risk Tobacco Product-related taxes) covering a broad range of tax magnitudes. Participants will complete two control trials and one tax proposal condition, with and without the conventional cigarettes available in the marketplace. Each condition (with and without conventional cigarettes) will include five price scenarios, with tax rates increasing across scenarios by a multiplicative factor. Tobacco products are placed into three tax tiers: high-, medium-, and no-tax, according to the goals of each proposal.

ELIGIBILITY:
Inclusion Criteria:

* provide informed consent
* provide a breath carbon monoxide sample ≥ 8 ppm,
* be at least 21 years of age (the legal age to purchase tobacco),
* smoke at least 10 cigarettes daily, and
* use other tobacco products less than weekly.

Exclusion Criteria:

* report uncontrolled physical or mental health conditions (e.g., uncontrolled diabetes, high blood pressure, major depressive disorder, etc.),
* use of smoking cessation medications (e.g., nicotine replacement, bupropion, varenicline) in the past 30 days,
* report concrete, immediate plans to alter/quit using their usual tobacco products in the next 30 days,
* be pregnant or lactating, or
* have plans to move out of the area during the experiment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percent of Budget Allocated to Products from each Tax Tier | Day 1
  The investigators will measure the percent of each participant's study budget spent on products from each of the three tax tiers (high-, medium, and no-tax).

SECONDARY OUTCOMES:
Quantity of Products Purchased from each Tax Tier | Day 1
  The investigators will measure the quantity of individual units of tobacco/nicotine products purchased from each tax tier (high-, medium, and no-tax).

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Stein, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC; Christine E Sheffer, Ph.D., Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Fralin Biomedical Research Institute at VTC, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No
The study team will share de-identified data upon request.